CLINICAL TRIAL: NCT03164642
Title: Enhancing Communication Between Children in EI and Their Depressed Mothers
Brief Title: Using the LENA System in Early Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Determined feasibility was needed before conducting this trial
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-2105a; 1R03HD086330-01 (NIH); 550KR141630 (Other Grant/Funding Number: NIH Clinical and Translational Science Award (CTSA))
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Depression
Keywords: Depressive Symptoms; Developmental Disabilities; Early Intervention; Language Development; Communication; Maternal Empowerment
MeSH Terms: conditions — Depression; Developmental Disabilities; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LENA with Feedback (Experimental): Mothers who will run the LENA system with their young children, AND who will receive feedback from their service providers on how to enhance the language the home language environment.
  Interventions: Behavioral: LENA with Feedback
- LENA no feedback (Placebo Comparator): Mothers who will only run the LENA system with their young children. These mothers will NOT receive feedback from their service providers on how to enhance the language the home language environment.
  Interventions: Behavioral: LENA no feedback

INTERVENTIONS:
Behavioral: LENA with Feedback — The LENA with Feedback intervention will involve mothers running the Language ENhancement Assessment/intervention system, an audiorecorder language pedometer that records adult speech centered on the child, child vocalizations, and parent-child reciprocal turn-taking conversations. During their regular EI providers will use a standardized feedback protocol that includes emphasizing the mother's strengths, reviewing the LENA visual output from the previous recording, and asking questions to elicit how the mother can increase her child-centered and reciprocal communications during daily routines. The conversation will include concrete examples of how the mother can increase the language exchanges, encouragement, and practical ways to individually tailor the strategies to the family.
  Arms: LENA with Feedback
Behavioral: LENA no feedback — The LENA with Feedback intervention will involve mothers running the Language ENhancement Assessment/intervention system, an audiorecorder language pedometer that records adult speech centered on the child, child vocalizations, and parent-child reciprocal turn-taking conversations
  Arms: LENA no feedback

SUMMARY:
This project will determine whether an intervention to enhance communication between infants and toddlers with developmental disabilities and their depressed mothers can be integrated into federally-funded Early Intervention (EI) services. Participants will be mothers with depressive symptoms whose children are receiving EI services, along with their EI service providers.

The investigators will conduct a small randomized control trial using the Language ENhancement Assessment/intervention system (LENA), a technology-supported language monitoring system, with 20 mothers and one of their child's EI service providers. The LENA uses an infant or toddler garment with an integrated audiotape system that records adult speech centered on the child, child vocalizations, and reciprocal parent-child turn-taking conversations. The LENA software produces visual feedback that a mother can use to focus her language interactions with her child. A "LENA with feedback" group will follow participants in the intervention over 5 weeks: 5 weeks of LENA data collection (with mothers running the system 1 day/week for 16 consecutive hours), with feedback during 3 weeks (baseline=LENA, no feedback; 3 week intervention=LENA with feedback; post-intervention=LENA, no feedback). A "LENA no feedback" group will complete LENA data collection at baseline on the same schedule but will not receive feedback. The main difference between groups will be provision of LENA feedback and strategies to promote increased mother-child interactions. This design allows the investigators to isolate the effect of LENA with feedback, and minimizes attributing changes in language environments due to exposure to LENA alone. The investigators will analyze data from measures on LENA communication data (adult word count, child vocalizations and conversational turn-taking), and measures of child language, maternal depressive symptoms, and child disability profiles.

DETAILED DESCRIPTION:
Early Intervention (EI) services are provided to infants and toddlers with documented developmental delays in all 50 states and US territories. EI improves long-term infant-toddler adaptation and lowers the cost of care if parents use the services. However, depressive symptoms can reduce mothers' ability to provide the daily child development-promoting activities recommended by EI, increasing the child's risk for communication and behavioral problems. Indeed, repeated studies have shown that depressive symptoms reduce mothers' consistent use of developmentally sensitive, child-centered speech which, in turn, lead to negative child cognitive and behavioral outcomes. Previous research showed that over one-third of mothers of children with disabilities have significant levels of depressive symptoms, a rate higher than the population at large. Infants and toddlers of depressed mothers have been shown to receive fewer intensive services and have been shown to interfere with uptake of EI services through impaired mother-child interactions. A preliminary study by the investigators found that over a third of mothers of infants and toddlers enrolled in EI in a large North Carolina county had severe depressive symptoms and depression histories. Fortunately, the investigators also found that when depressed mothers were provided with concrete, attainable skills for improving interactions with their child, the impact of depression on both mother and child was substantially reduced. Focusing on a depressed mother's child-centered speech and reciprocal communication also improves child outcomes, even when the child is cognitively compromised. However, none of these specialized services are part of EI best practices. Thus, EI is an ideal setting in which to integrate screening, referral and targeted skills for depressed mothers in order to improve parent-child interactions and ultimately, child outcomes.

This project will develop an intervention focused on communication between infants and toddlers with diagnosed or suspected developmental disabilities and their mothers who have depressive symptoms. The primary aim of the study is to test the initial efficacy of embedding a language pedometer, the Language ENhancement Assessment/intervention system (LENA), into EI to teach mothers to increase child-centered speech and reciprocal communication, which have been linked to positive child outcomes, and to increase parenting efficacy in depressed mothers of children in EI. While maternal depressive symptoms can disrupt developmentally stimulating, child-centered speech, simple tools to assess and provide feedback to mothers can improve the child-centered speech and reciprocal language interactions that positively impact child outcomes. Although the LENA has been used in other studies and shown improvements in mothers' child-centered speech, the system has not been used with mothers showing depressive symptoms or in the EI context.

Using a randomized wait-list controlled design, the investigators will examine whether use of the LENA with feedback from a supportive EI provider has an impact on the child's language environment, parenting efficacy and maternal depressive symptoms. The investigators will stratify mothers by group based on depressive symptoms (mild, moderate, moderately severe) and randomly assign them to intervention (LENA with feedback) or wait-list control (LENA no feedback). The investigators will examine the use of the LENA system and the impact on short term child outcomes including receptive/expressive language, functional and social communication, and social-emotional behavior, and on maternal depressive symptoms. Positive intervention outcomes may ultimately lead to a sustainable addition to EI programs in all 50 US states and territories.

ELIGIBILITY:
Inclusion Criteria:

Service Coordinator and Service Provider Inclusion:

* Be a CDSA employee in Durham, Wake, Alamance or Guilford Counties, NC
* Be a service coordinators or approved Speech-Language Provider(SLP) or Community Based Rehabilitative Service (CBRS) provider (service providers).
* Eligibility of the service providers will be determined by the agreement of a mother to participate in the LENA portion of the study and the agreement of the service providers to participate as well.

Mothers Inclusion criteria:

* Be 18 years or older. Mothers who are 18 years can give consent independently.
* Be the biological or adoptive mother of an infant (6 weeks - 18 months old) or toddler (19 -32 months old) enrolled in EI at the time of recruitment; mothers must be the primary caretaker of the child.
* EI services are offered only to infants and toddlers up to the age of 36 months; this study caps the age of enrollment at 32 months to ensure that toddlers are continuously enrolled in EI during the data collection period.
* Able to independently give consent. Mothers must have adequate capacity to participate in the LENA intervention as well as understand what they will be asked to do as participants.
* Score 8 or higher on the PHQ-9. This score is indicative of depressive symptoms.

Exclusion Criteria:

Service Coordinator and Service Provider Inclusion: none

Mothers Exclusion criteria:

* Currently pregnant by self-report.
* Child is completely deaf

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in LENA Adult Word Count score after 5 weeks | pre/post for a 5-week intervention window
  The LENA system, which records adult-child vocalizations, measures the number of the target adult's (e.g., parent) child-directed words (child-directed speech). The total possible range is 0-n, where higher scores indicate an increased number of child-directed words spoken by the target adult and higher degrees of a language-rich environment. Lower scores indicate fewer words spoken by the target adult and represent an environment that is not language-rich.

SECONDARY OUTCOMES:
Change in Parenting Sense of Competence Scale Efficacy subscale score after 5 weeks | pre/post for a 5-week intervention window
  The Parenting Sense of Competence Scale is a 17-item measure assessing parental competence. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". The Efficacy subscale measures feelings of efficacy as a parent. It has 7 questions (1,6,7,10,11,13,15), producing a range of 6-42. Higher scores indicate greater self-efficacy. Lower scores mean more impairment.
Change in Patient Health Questionnaire-9 (PHQ-9) score after 5 weeks | pre/post for a 5-week intervention window
  The PHQ-9 is a depression scale used to assess brief depression severity by rating symptoms and functional impairment experienced in the last two weeks. The questionnaire contains a total of 9 questions, and each question is scored on a range from 0-3. The minimum value "0" represents not at all, "1" several days, "2" indicates more than half the days, and the maximum value "3" stands for nearly every day. The total possible range is 0-27, with higher scores indicating more depressive symptoms. The total number of each 0, 1, 2, 3 is added and multiplied by its value (0=0, 1=1, etc.) to produce a total score generated from the subtotal sum. The PHQ-9 total score is interpreted as follows: 0-4 represents minimal depression, 5-9 as mild depression, 10-14 as moderate depression, 15-19 moderately severe depression, and 20-27 severe depression.
Change in LENA Mother/Child Turn-Taking score after 5 weeks | pre/post for a 5-week intervention window
  The LENA system, which records adult-child vocalizations, measures the number of conversational turns between the target adult (e.g., parent) and child. The total possible range is 0-n, where higher scores indicate an increased number of turns (back-and-forth, or "reciprocal" language exchanges) between the adult and child, reflecting higher degrees of a language-rich environment. Lower scores indicate fewer conversational turns between the adult and child, and represent an environment that is not language-rich.
Change in LENA Child Vocalization score after 5 weeks | pre/post for a 5-week intervention window
  The LENA system, which records adult-child vocalizations, measures the number of vocalizations of the target child. The total possible range is 0-n, where higher scores indicate an increased number of vocalizations from the child, reflecting higher levels of language development. Lower scores indicate fewer vocalizations from child, and represent lower levels of language development.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Beeber, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Anne Wheeler, PhD, Principal Investigator — RTI International; Doré LaForett, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Durham Children's Developmental Services Agency, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No